CLINICAL TRIAL: NCT01776060
Title: Serial Collection of Primary Progressive Multiple Sclerosis Participants in the MURDOCK Study
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00040961
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Primary Progressive Multiple Sclerosis
Keywords: Primary Progressive Multiple Sclerosis; Multiple Sclerosis; biomarker; 'omic; progression
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood (RNA/DNA), serum, plasma, urine
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: generation of 'omic markers of disease progression — Aside from first in disease sampling, the serial, biannual collection of samples from PPMS patients would not only permit the identification of 'omic profiles that can be compared and contrasted to those from RRMS patients in a parallel study, but it would also allow the generation of 'omic markers of disease progression.

SUMMARY:
The goal of this study is to enroll 100 participants with Primary Progressive Multiple Sclerosis (PPMS) that have joined the MURDOCK Study Horizon 1.5 (Duke IRB Pro00011196) and the Multiple Sclerosis cohort (Duke IRB Pro00023791). All 100 participants will complete a biannual collection of a follow up questionnaire and blood/urine collection for a period of 5 years.

DETAILED DESCRIPTION:
Unlike Relapsing Remitting Multiple Sclerosis (RRMS) or Secondary Progressive Multiple Sclerosis (SPMS) in which patients experience a remission or lessening of their symptoms, Primary Progressive Multiple Sclerosis (PPMS) is characterized by progression of disability from onset, with no, or only occasional and minor, remissions and improvements. The age of onset for the primary progressive subtype is later than for the relapsing-remitting, but similar to mean the age of progression between the relapsing-remitting and the secondary progressive - around 40 years of age. Because of its prevalence, RRMS represents the largest basis for basic and clinical MS research. Therefore, drugs have primarily been developed to slow disease progression in RRMS and SPMS patients. No treatment has been proven successful in treating primary progressive MS.

The MURDOCK-MS collection represents a unique opportunity to carry out detailed biomarker research on PPMS patients and, to the knowledge of this investigator and his colleagues in the field, would represent an exceptional cohort that is not available elsewhere in the US or the rest of the world. Aside from first in disease sampling, the serial, biannual collection of samples from PPMS patients would not only permit the identification of 'omic profiles that can be compared and contrasted to those from RRMS patients in a parallel study, but it would also allow the generation of 'omic markers of disease progression. This progressive etiology would provide valuable insight into PPMS development and may also shed light on SPMS progression.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the MURDOCK Study Horizon 1.5 (Pro00011196)
* Enrolled in the Multiple Sclerosis Cohort (Pro00023791)
* Diagnosed with Primary Progressive Multiple Sclerosis
* At least 18 years of age

Exclusion Criteria:

* Participants not willing to participate or sign informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must enroll in the MURDOCK Study Horizon 1.5 (Pro00011196) as well as the Multiple Sclerosis cohort (Pro00023791) in order to participate in this biannual collection of a follow up questionnaire and blood/urine collection for participants who have Primary Progressive MS. The biannual collection will continue for 5 years. Those participants with PPMS who are already enrolled in the MURDOCK Study Horizon 1.5 and Multiple Sclerosis cohort will be contacted via phone to assess interest in the PPMS study. New participants with PPMS who enroll into the Horizon 1.5 study and Multiple Sclerosis cohort will be asked during the time of enrollment if they would like to participate in the PPMS study as well.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
Generation of 'omic markers of disease progression | 5 years
  Biannual collection of samples from PPMS patients would not only permit the identification of 'omic profiles that can be compared and contrasted to those from RRMS patients in a parallel study, but it would also allow the generation of 'omic markers of disease progression. This progressive etiology would provide valuable insight into PPMS development and may also shed light on SPMS progression.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Gr, PhD, Principal Investigator — Duke Medicine Site Based Research Group
Locations (3):
- United States (3):
  - NE Neurology, Concord, North Carolina
  - The Stedman Center on the Duke Center for Living Campus, Durham, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina

REFERENCES:
- See also: Related Info — http://www.murdock-study.com